CLINICAL TRIAL: NCT06577532
Title: A Clinical Study to Investigate Safety, Tolerability, Immunogenicity, and Preliminary Efficacy of mRNA Nanoparticles Encoding KRAS Neoantigens (ABO2102) in Participants With KRAS-mutated Advanced Pancreatic Cancer And Other Solid Tumors
Brief Title: Study of KRAS Neoantigen mRNA Vaccine (ABO2102) in Patients With KRAS -Mutated Solid Tumors
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Suzhou Abogen Biosciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ABO2102-001
Record Dates: First submitted 2024-08-22; First posted 2024-08-29 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Pancreatic Neoplasms; Other Solid Tumors
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ABO2102 (Experimental): Prat I: Monotherapy
  Interventions: Drug: ABO2102
- ABO2102 and Toripalimab (Experimental): Part I&II: ABO2102 in combination with Toripalimab
  Interventions: Drug: ABO2102; Drug: Toripalimab

INTERVENTIONS:
Drug: ABO2102 — mRNA encoding mutant KRAS neoantigens, administrated intramuscularly
Drug: Toripalimab — Anti-PD-1 antibody, administered intravenously
  Arms: ABO2102 and Toripalimab

SUMMARY:
The purpose of this study is to evaluate the safety, immunogenicity, pharmacodynamics, as well as preliminary efficacy of KRAS neoantigen mRNA vaccine (ABO2102) alone and in combination with toripalimab (anti-PD-1 monoclonal antibody) among participants with KRAS-mutated advanced pancreatic cancer and other solid tumors. The trial includes dose escalation (Part I) and dose expansion(Part II) parts.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age at time of informed consent.
2. Participants with histologically and/ or cytologically confirmed advanced solid tumors (such as pancreatic ductal adenocarcinoma, non-small cell lung cancer, etc.), whose disease has progressed or being intolerant to relevant treatments during or following at least one line of systemic treatment; patients in the second stage include those who have experienced disease progression or intolerance to previous systemic treatments, as well as those who have not received systemic therapy but are deemed by the investigator to potentially benefit from the study treatment based on a comprehensive clinical assessment.
3. Harboring at least one of the targeted KRAS mutants.
4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0~2.
5. Life expectancy of ≥12 weeks.
6. Sufficient organ function.

Exclusion Criteria:

1. Any other prior malignancy active within the previous 5 years, except for skin basal cell cancer that have been cured, superficial bladder cancer, or carcinoma in situ of the breast or cervix.
2. Received KRAS cancer vaccine before.
3. Immunosuppressants or other immunomodulatory drugs were required within 4 weeks before the first dose of study treatment. Physiological doses of systemic steroids or topical medications are allowed. Topical medications should not exceed the dose recommended in the package insert or have any systemic exposure signs; Or patients with other acquired or congenital immunodeficiency diseases, or a history of organ transplantation who need to use immunosuppressants or other immunomodulatory drugs.
4. History of severe allergies or known allergies to any active or inactive component of the study drug(s).
5. Uncontrolled systemic infection; active tuberculosis.
6. Severe cardiovascular diseases.
7. Has known symptomatic, untreated central nervous system metastases, or CNS metastases requiring continued treatment. Participants with asymptomatic brain metastases and who do not require treatment are eligible for enrolment.
8. Have active autoimmune and inflammatory diseases.
9. Have immediate hypersensitivity, a history of eczema or asthma uncontrolled by topical corticosteroids.
10. Have other serious medical conditions
11. A history of organ transplantation, bone marrow transplantation or hematopoietic stem cell transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Part I: The incidence and nature of dose-limiting toxicity (DLT) for ABO2102 as monotherapy or in combination with toripalilmab. | 21 days after the first dose of study treatment
Part I: The incidence and severity of treatment-emergent adverse events (TEAE)s. | from the first dose of study treatment to 30 days after the last dose of monotherapy or to 90 days after the last dose of the combination therapy.
Part I: The incidence and severity of serious TEAEs (TESAE)s. | from the first dose of study treatment to 30 days after the last dose of monotherapy or to 90 days after the last dose of the combination therapy.
Part I: The incidence and severity of TEAEs leading to interruption or early termination of study treatment. | from the first dose of study treatment to 30 days after the last dose of monotherapy or to 90 days after the last dose of the combination therapy.
Part II: Overall Response Rate (ORR) per RECIST version 1.1. | from the first dose of study treatment to up to 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Baiyong Shen, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No